CLINICAL TRIAL: NCT04591418
Title: Farklı çürük Temizleme yöntemlerinin çocuk Hastalarda Klinik Olarak karşılaştırılması
Brief Title: A Comparative Clinical Study of Different Caries Removal Techniques in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, volkan Ciftci, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 94/57
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries in Children
Keywords: Er:YAG laser; Caries removal; Dental anxiety; Acceptability
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotary handpieces (Active Comparator)
  Interventions: Device: Rotary handpieces
- Er:YAG laser (Experimental)
  Interventions: Device: Er:YAG laser

INTERVENTIONS:
Device: Rotary handpieces — Dental Caries removal
  Arms: Rotary handpieces
Device: Er:YAG laser — Dental Caries removal
  Arms: Er:YAG laser

SUMMARY:
The aim of this study is to evaluate the acceptance of pediatric patiens using Er: YAG laser in comparison with the conventional techniques for caries removal.

The study was carried out on 100 children between the ages of 9-12, who had class 1 occlusal caries in one of their permanent first molars. The patients were divided into two groups; conventional technical group and laser group. Rotary handpieces was used in conventional technique group, Er:YAG laser was used in the laser group for caries removal. The heart rate of each patient was measured during the caries removal procedure at 30 seconds intervals. The pain during the procedure was determined by VAS. CFSS-DS scale was used to determine the anxiety level of the patients before and after the procedure. FIS was used to determine how patients are disturbed from the smell, taste, sound, vibration and sight of the devices after the procedure. The video segments were collected from the patients during the caries removal and the procedural pain were evaluated by the FLACC scale.

DETAILED DESCRIPTION:
Based our results, ın the laser group, the patients were found to experience less pain and discomfort compared to conventional technique according to the VAS and FLACC scores. The rate of patients with dental anxiety decreased significantly in the laser group compared with the conventional group according to CFSS-DS performed after the procedure. According to the sensory survey, the laser group had good acceptability compared to the conventional technique group in terms of vibration and sight. The laser group showed a lower percentage increase in heart rate comparsion between beginning and end of procedure. It was observed that the cavity preparation time was longer in the laser group.

ELIGIBILITY:
Inclusion Criteria:

* patients age between 9-12 years old
* Having no systemic condition and ASA 1 healty status
* Having lower permanent first molar teeth with occlusal caries (class 1)
* having no laser treatment before

Exclusion Criteria:

* having spontaneous tooth pain
* having high dental anxiety
* having no restorative treatment before
* teeth with periapical pathology, a root filling or non-vital teeth.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Comfort | through study completion, an average of 6 months
  Units on a Scale ( Patient comfort was evaluated with Facial Image Scale after treatment. Patients signed from 1 to 5 score for treatment comfort.The data were collected and statistically analysed using by the numerical data. In this study, "1" and "2" scores are considered as better outcome. Patients who signed these scores described as good comfortable. The worst outcome is considered as the patients signed "4-5". Each scale range for each time interval evaluated as count of patient and presented as percentage.)
Dental anxiety | through study completion, an average of 6 months
  Units on a Scale (Dental anxiety was evaluated with Dental Subscale of the Children's Fear Survey Schedule after treatment. The patients signed from 0 to 38 score for dental anxiety after the treatment.The data were collected and statistically analysed using by the numerical data. In this study, " 0-38" scores are considered as better outcome. Patients who were have these scores described no dental anxiety for treatment. The worst outcome is considered as the patients have ">38". Each scale range for each time interval evaluated as count of patient and presented as percentage.)
Changes in pain | through study completion, an average of 6 months
  Units on a Scale (Changes in pain was evaluated with Legs, Activity, Cry, Consolability scale after treatment. Observer signed from 0 to 3 score for treatment pain during the treatment.The data were collected and statistically analysed using by the numerical data. In this study, "0" and "1" scores are considered as better outcome. Patients who were signed these scores described as no pain for treatment. The worst outcome is considered as the patients signed "2-3". Each scale range for each time interval evaluated as count of patient and presented as percentage.)

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)